CLINICAL TRIAL: NCT05097287
Title: A Randomized, Double-Blind, Placebo Controlled Study Assessing the Long-term Effect of Dupilumab on Prevention of Lung Function Decline in Patients With Uncontrolled Moderate to Severe Asthma
Brief Title: Study Assessing the Long-term Effect of Dupilumab on Prevention of Lung Function Decline in Adult Patients With Uncontrolled Moderate to Severe Asthma
Acronym: ATLAS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPS16676; U1111-1266-2849 (Registry Identifier: ICTRP); 2024-513423-16 (Registry Identifier: CTIS); 2021-003903-16 (EudraCT Number)
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab (Experimental): Dupilumab administered every 2 weeks (Q2W) after an initial loading dose (2 injections) on Day 1
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Matching placebo administered Q2W after an initial loading dose (2 injections) on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — solution for injection subcutaneous
  Arms: Dupilumab
Drug: Placebo — solution for injection subcutaneous
  Arms: Placebo

SUMMARY:
This is an interventional, randomized, parallel group, treatment, Phase 3b/4, double blind, 2-arm study to assess the effect of dupilumab compared to standard of care therapy on preventing or slowing the rate of lung function decline in adult patients with uncontrolled moderate to severe asthma.

The estimated duration is 4±1 weeks of screening and run-in period, followed by a 3-year double blinded treatment period. There will be a post-treatment follow-up (FU) period up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 (or the legal age of consent in the jurisdiction in which the study is taking place) years of age inclusive, at the time of signing the informed consent.
* Patients with a physician diagnosis of asthma (according to Global Initiative for Asthma (GINA) 2021) for ≥12 months
* Treatment with medium to high dose inhaled corticosteroids (ICS) in combination with a second controller (eg, long-acting beta-2 adrenergic receptor agonists (LABA), leukotriene receptor antagonists (LTRA) with a stable dose ≥1 month prior to Visit 1. Patients requiring a third controller for their asthma will be considered eligible for this study, and it should also be on stable dose ≥1 month prior to Visit 1. Patients requiring an additional controller as a fourth controller (Montelukast) for another type 2 comorbid condition such as allergic rhinitis will be considered eligible for this study, and should be on a stable dose for ≥1 month prior to Visit 1.
* Pre-bronchodilator forced expiratory volume (FEV1) ≤ 80% of predicted normal for adults at Visits 1 and 2, prior to randomization
* Asthma Control Questionnaire 5-question version (ACQ-5) score ≥1.5 at Visits 1 and 2, prior to randomization.
* Variable airflow obstruction as documented by one or more of the following (at least 1 needs to be met):

  i) Positive reversibility test: ≥12% and 200 mL improvement in FEV1 after SABA administration prior to randomization, or documented in the 24 months prior to Visit 1. OR, ii) Positive bronchial challenge test: fall in FEV1 of ≥20% with standard doses of methacholine, or ≥15% with standardized hyperventilation, hypertonic saline or mannitol challenge prior to randomization or documented in the 24 months prior to Visit 1 OR, iii) Average daily diurnal Peak flow variability of >10% over a 2-week period, documented in the past 24 months prior to Screening Visit 1. OR, iv) Airflow variability in clinic FEV1 >12% and 200 mL between visits outside of respiratory infections, documented in the past 24 months prior to Screening Visit 1. OR v) FEV1 increases by more than 12% and 200mL from baseline after 4 weeks of anti-inflammatory treatment.
* Reversibility test: Three attempts may be made during the Screening Period until the Baseline visit to meet the qualifying criteria for reversibility. This is only required if reversibility or other evidence of expiratory airflow limitation eligibility criteria was not performed within 24 months prior to Visit 1.
* FeNO ≥35 ppb at Visit 2, prior to randomization.
* History of ≥1 severe exacerbation(s) in the previous year before Visit1 defined as a deterioration of asthma requiring:

  i) Use of systemic corticosteroids for ≥3 days; or ii) Hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* History or clinical evidence of chronic obstructive pulmonary disease (COPD) including Asthma-COPD Overlap Syndrome (ACOS) or any other significant lung disease (eg, emphysema, lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, Churg-Strauss Syndrome).
* Severe asthma exacerbation requiring treatment with systemic corticosteroid (SCS) in the past month before visit 1 or during the screening period.
* Current acute bronchospasm or status asthmaticus.
* Diagnosed pulmonary (other than asthma) or systemic disease associated with elevated peripheral eosinophil counts.
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study. Examples include, but are not limited to, participants with short life expectancy, uncontrolled diabetes, cardiovascular conditions, severe renal conditions (eg, participants on dialysis), or other severe endocrinological, gastrointestinal, metabolic, pulmonary, psychiatric, or lymphatic diseases. The specific justification for participants excluded under this criterion will be noted in the study documents (chart notes, case report forms [CRFs], etc).
* Patients with active tuberculosis (TB) or non-tuberculous mycobacterial infection, or a history of incompletely treated TB will be excluded from the study unless it is well documented by a specialist that the participant has been adequately treated and can now start treatment with a biologic agent, in the medical judgment of the Investigator and/or infectious disease specialist. Tuberculosis testing will be performed on a country by country basis, according to local guidelines if required by regulatory authorities or ethics boards, or if TB is suspected by the investigator
* Known or suspected immunodeficiency, including history of invasive opportunistic infections (eg, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency or prolonged duration suggesting an immune-compromised status, as judged by the Investigator.
* Active malignancy or history of malignancy within 5 years before Visit 1 (screening visit), except completely treated in situ carcinoma of the cervix and completely treated and resolved non metastatic squamous or basal cell carcinoma of the skin.
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antifungals or receiving only symptomatic treatment (e.g. influenza or COVID-19) within 2 weeks before the screening visit (Visit 1) or during the screening period.
* History of human immunodeficiency virus (HIV) infection or positive HIV 1/2 serology at Visit 1 (screening visit).
* Diagnosed with, suspected of, or at high risk of endoparasitic infection, and/or use of antiparasitic drugs within 2 weeks before Visit 1 (screening visit) or during the screening and run-in period
* Current smoker (cigarette or e-cigarette) or cessation of smoking within 6 months prior to Visit 1.
* Previous smoker with a smoking history >10 pack-years.
* History of systemic hypersensitivity or anaphylaxis to dupilumab or any other biologic therapy, including any excipient.
* Any biologic therapy (including experimental treatments and dupilumab) or any other biologic therapy/immunosuppressant/immunomodulators within 4 weeks prior to V1 or 5 half-lives, whichever is longer.
* Treatment with a live (attenuated) vaccine within 4 weeks before Visit 1 (screening visit) or during the screening period.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1324 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-08-21 (Estimated)

PRIMARY OUTCOMES:
Rate of change from week 8 to week 52 on post-BD FEV1 slope in FeNO population | Week 8 to Week 52
  Rate of change from week 8 to week 52 on post-bronchodilator (BD) forced expiratory volume in one second (FEV1) slope in FeNO population.

SECONDARY OUTCOMES:
Rate of change from week 8 to week 52 on post-BD FEV1 slope in the Total population | Week 8 to Week 52
  Rate of change from week 8 to week 52 on post-BD FEV1 slope in the Total population.
Rate of change from week 8 to week 104 on post-BD FEV1 slope in the FeNO population | Week 8 to Week 104
  Rate of change from week 8 to week 104 on post-BD FEV1 slope in the FeNO population.
Change from baseline to week 52 in pre-BD FEV1 in FeNO and Total populations | Baseline to Week 52
  Change from baseline to week 52 in pre-BD FEV1 in FeNO and Total populations.
Change from baseline to week 52 in post-BD FEV1 in FeNO and Total populations | Baseline to Week 52
  Change from baseline to week 52 in post-BD FEV1 in FeNO and Total populations.
Annualized severe exacerbation rate during the 52-week period in FeNO and Total populations | Baseline to Week 52
  Exacerbation defined as a deterioration of asthma requiring use of systemic corticosteroids for ≥3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids.
Change from baseline to week 52 in fractional exhaled nitric oxide (FeNO) levels in FeNO and Total populations | Baseline to Week 52
  Change from baseline to week 52 in FeNO levels in FeNO and Total populations.
Change from baseline to week 52 in Asthma Control Questionnaire 7 items (ACQ-7) in FeNO and Total populations | Baseline to Week 52
  ACQ-7 was designed to measure both the adequacy of asthma control and change in asthma control. A global score ranges between 0 (totally controlled) and 6 (severely uncontrolled). Higher score indicates lower asthma control.
Change from baseline to week 52 in pre-BD FEV1 % predicted in FeNO and Total populations | Baseline to Week 52
  Change from baseline to week 52 in pre-BD FEV1 % predicted in FeNO and Total populations.
Change from baseline to week 52 in Forced Vital Capacity (FVC) in FeNO and Total populations | Baseline to Week 52
  Change from baseline to week 52 in FVC in FeNO and Total populations.
Rate of change from week 8 to week 104 on post-BD FEV1 slope in Total Population | Week 8 to Week 104
  Rate of change from week 8 to week 104 on post-BD FEV1 slope in Total Population.
Change from baseline to week 104 in pre-BD FEV1 in FeNO and Total populations | Baseline to Week 104
  Change from baseline to week 104 in pre-BD FEV1 in FeNO and Total populations.
Change from baseline to week 104 in post-BD FEV1 in FeNO and Total populations | Baseline to Week 104
  Change from baseline to week 104 in post-BD FEV1 in FeNO and Total populations.
Annualized severe exacerbation rate during the 104-week period in FeNO and Total populations | Baseline to Week 104
  Exacerbation defined as a deterioration of asthma requiring use of systemic corticosteroids for ≥3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids.
Change from baseline to week 104 in FeNO levels in FeNO and Total populations | Baseline to Week 104
  Change from baseline to week 104 in FeNO levels in FeNO and Total populations.
Change from baseline to week 104 in ACQ-7 in FeNO and Total populations | Baseline to Week 104
  ACQ-7 was designed to measure both the adequacy of asthma control and change in asthma control. A global score ranges between 0 (totally controlled) and 6 (severely uncontrolled). Higher score indicates lower asthma control.
Change from baseline to week 104 in pre-BD FEV1 % predicted in FeNO and Total populations | Baseline to Week 104
  Change from baseline to week 104 in pre-BD FEV1 % predicted in FeNO and Total populations.
Change from baseline to week 104 FVC in FeNO and Total populations | Baseline to Week 104
  Change from baseline to week 104 FVC in FeNO and Total populations.
Change from baseline to week 52 in Asthma Quality Of Life Questionnaire with Standardized Activities (AQLQ(S)) in FeNO and Total populations | Baseline to Week 52
  The AQLQ (S) was designed as a self-administered patient reported outcome to measure the functional impairments that are most troublesome to patients as a result of their asthma. A global score is calculated ranging from 1 to 7. Higher scores indicate better quality of life.
Change from baseline to week 104 in AQLQ(S) in FeNO and Total populations | Baseline to Week 104
  The AQLQ (S) was designed as a self-administered patient reported outcome to measure the functional impairments that are most troublesome to patients as a result of their asthma. A global score is calculated ranging from 1 to 7. Higher scores indicate better quality of life.
Rate of change from week 8 to week 156 on post-BD FEV1 slope in FeNO and Total populations | Week 8 to Week 156
  Rate of change from week 8 to week 156 on post-BD FEV1 slope in FeNO and Total populations.
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline to Week 168
  Incidence of TEAEs and SAEs.
Incidence of adverse events of special interest (AESIs) | Baseline to Week 168
  Incidence of AESIs.

CONTACTS AND LOCATIONS:
Locations (249):
- United States (74):
  - Cullman Research Center- Site Number : 8400001, Cullman, Alabama
  - Shoals Primary Care - Sheffield- Site Number : 8400015, Sheffield, Alabama
  - Chandler Clinical Research Trials- Site Number : 8400147, Chandler, Arizona
  - Pulmonary Associates - Deer Valley Office- Site Number : 8400155, Phoenix, Arizona
  - Medical Advancement Center of Arizona (MACOA)- Site Number : 8400130, Tempe, Arizona
  - Del Sol Research Management - Tucson- Site Number : 8400017, Tucson, Arizona
  - Kern Allergy and Medical Research- Site Number : 8400037, Bakersfield, California
  - Vitality Clinical Research- Site Number : 8400142, Beverly Hills, California
  - ASCADA Research- Site Number : 8400076, Fullerton, California
  - Allergy and Asthma Specialists Medical Group- Site Number : 8400162, Huntington Beach, California
  - Newport Native MD- Site Number : 8400054, Newport Beach, California
  - Prospective Research Innovations- Site Number : 8400131, Rancho Cucamonga, California
  - Mercy Medical Group - Midtown- Site Number : 8400164, Sacramento, California
  - Integrated Research of Inland- Site Number : 8400156, Upland, California
  - Allianz Research Institute- Site Number : 8400018, Westminster, California
  - Woodland Clinic - Woodland- Site Number : 8400171, Woodland, California
  - Central Florida Pulmonary Group - Altamonte Springs- Site Number : 8400035, Altamonte Springs, Florida
  - Florida Center for Allergy & Asthma Research- Site Number : 8400032, Aventura, Florida
  - Beautiful Minds Clinical Research Center- Site Number : 8400141, Cutler Bay, Florida
  - Omega Research Consultants - Debary - North Charles Richard Beall Boulevard- Site Number : 8400023, DeBary, Florida
  - Florida Lung, Asthma and Sleep Specialists (FLASS) - Polynesian- Site Number : 8400098, Kissimmee, Florida
  - Ivetmar Medical Group- Site Number : 8400063, Miami, Florida
  - My Preferred Research- Site Number : 8400073, Miami, Florida
  - Research Institute of South Florida- Site Number : 8400079, Miami, Florida
  - Floridian Clinical Research - Miami Lakes- Site Number : 8400091, Miami Lakes, Florida
  - Heuer M.D. Research- Site Number : 8400024, Orlando, Florida
  - JSV Clinical Research- Site Number : 8400150, Tampa, Florida
  - Appalachian Clinical Research- Site Number : 8400129, Adairsville, Georgia
  - Alpha Clinical Research Group - Dunwoody- Site Number : 8400116, Dunwoody, Georgia
  - Aeroallergy Research Laboratory- Site Number : 8400114, Savannah, Georgia
  - Rush University Medical Center- Site Number : 8400146, Chicago, Illinois
  - NorthShore University Health System - Endeavor Health Medical Group - Skokie - Woods Drive- Site Number : 8400138, Skokie, Illinois
  - Family Allergy & Asthma - Louisville - Goss Avenue- Site Number : 8400160, Louisville, Kentucky
  - Allergy and Asthma Specialist- Site Number : 8400007, Owensboro, Kentucky
  - Avant Research Associates - Crowley- Site Number : 8400117, Crowley, Louisiana
  - Tandem Clinical Research - Metairie- Site Number : 8400163, Metairie, Louisiana
  - Javara Privia Mid-Atlantic - Annapolis- Site Number : 8400087, Annapolis, Maryland
  - Urgent Care Clinical Trials and KUR Research- Site Number : 8400169, Columbia, Maryland
  - Chesapeake Clinical Research - White Marsh- Site Number : 8400119, White Marsh, Maryland
  - Genesis Clinical Research - Fall River- Site Number : 8400050, Fall River, Massachusetts
  - University of Michigan Health System - Ann Arbor- Site Number : 8400030, Ann Arbor, Michigan
  - Revival Research Institute - Dearborn- Site Number : 8400097, Dearborn, Michigan
  - Revive Research Institute- Site Number : 8400100, Lathrup Village, Michigan
  - Romedica- Site Number : 8400043, Rochester, Michigan
  - Great Lakes Research Institute Site Number : 8400111, Southfield, Michigan
  - Great Lakes Research Institute - Southfield- Site Number : 8400111, Southfield, Michigan
  - Allergy & Immunology Associates of Ann Arbor- Site Number : 8400107, Ypsilanti, Michigan
  - The Asthma and Allergy Center- Site Number : 8400055, Bellevue, Nebraska
  - Jersey City Breathing Center: Elamir Mazhar- Site Number : 8400143, Jersey City, New Jersey
  - Urban Health Plan- Site Number : 8400144, The Bronx, New York
  - Clinical Research Of Gastonia- Site Number : 8400012, Gastonia, North Carolina
  - Advanced Respiratory and Sleep Medicine - Huntersville- Site Number : 8400056, Huntersville, North Carolina
  - Lapis Clinical Research - Mooresville- Site Number : 8400112, Mooresville, North Carolina
  - Southeastern Research Center- Site Number : 8400153, Winston-Salem, North Carolina
  - Asthma & Allergy Center - Toledo- Site Number : 8400051, Toledo, Ohio
  - St. Luke's University Hospital- Site Number : 8400099, Bethlehem, Pennsylvania
  - Temple University Hospital- Site Number : 8400038, Philadelphia, Pennsylvania
  - Allergy & Clinical Immunology Associates Pittsburgh- Site Number : 8400042, Pittsburgh, Pennsylvania
  - Bogan Sleep Consultants- Site Number : 8400102, Columbia, South Carolina
  - ADAC Research- Site Number : 8400026, Greenville, South Carolina
  - Main Street Physician's Care- Site Number : 8400077, Little River, South Carolina
  - National Allergy and Asthma - North Charleston - Northside Drive- Site Number : 8400092, North Charleston, South Carolina
  - Health Concepts- Site Number : 8400006, Rapid City, South Dakota
  - REX Clinical Trials - Beaumont- Site Number : 8400135, Beaumont, Texas
  - South Texas Medical Research Institute - TTS Research- Site Number : 8400009, Boerne, Texas
  - Discovery Clinical Trials - Dallas- Site Number : 8400123, Dallas, Texas
  - IntraCare- Site Number : 8400003, Dallas, Texas
  - C & R Research Services - Houston- Site Number : 8400067, Houston, Texas
  - Clear Brook Medical Associates- Site Number : 8400080, Houston, Texas
  - Metroplex Pulmonary and Sleep Center- Site Number : 8400014, McKinney, Texas
  - Andante Research- Site Number : 8400140, San Antonio, Texas
  - DM Clinical Research - 710 Lawrence Street- Site Number : 8400103, Tomball, Texas
  - Burke Internal Medicine and Research- Site Number : 8400170, Burke, Virginia
  - University of Virginia- Site Number : 8400082, Charlottesville, Virginia
- Belgium (2):
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560003, Liège
- Brazil (9):
  - Associacao Proar- Site Number : 0760004, Salvador, Estado de Bahia
  - Santa Casa de Misericordia de Belo Horizonte- Site Number : 0760006, Belo Horizonte, Minas Gerais
  - Health & Care - Consultancy, Research and HealthCare Management- Site Number : 0760010, Belém, Pará
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760003, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão- Site Number : 0760002, Blumenau, Santa Catarina
  - Clinica de Alergia Martti Antila- Site Number : 0760009, Sorocaba, São Paulo
  - Hospital Alemao Oswaldo Cruz - São Paulo- Site Number : 0760007, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 0760008, São Paulo
- Bulgaria (8):
  - Investigational Site Number : 1000005, Dupnitsa
  - Investigational Site Number : 1000012, Plovdiv
  - Investigational Site Number : 1000011, Rousse
  - Investigational Site Number : 1000002, Sofia
  - Investigational Site Number : 1000008, Sofia
  - Investigational Site Number : 1000009, Sofia
  - Investigational Site Number : 1000014, Sofia
  - Investigational Site Number : 1000013, Vratsa
- Canada (17):
  - Investigational Site Number : 1240028, Calgary, Alberta
  - Investigational Site Number : 1240020, Kelowna, British Columbia
  - Investigational Site Number : 1240022, Vancouver, British Columbia
  - Investigational Site Number : 1240004, Vancouver, British Columbia
  - Investigational Site Number : 1240010, Moncton, New Brunswick
  - Investigational Site Number : 1240015, Ajax, Ontario
  - Investigational Site Number : 1240018, Niagara Falls, Ontario
  - Investigational Site Number : 1240011, Toronto, Ontario
  - Investigational Site Number : 1240001, Toronto, Ontario
  - Investigational Site Number : 1240007, Toronto, Ontario
  - Investigational Site Number : 1240003, Windsor, Ontario
  - Investigational Site Number : 1240014, Montreal, Quebec
  - Investigational Site Number : 1240017, Montreal, Quebec
  - Investigational Site Number : 1240023, Montreal, Quebec
  - Investigational Site Number : 1240002, Québec, Quebec
  - Investigational Site Number : 1240025, Sherbrooke, Quebec
  - Investigational Site Number : 1240024, Saskatoon, Saskatchewan
- China (25):
  - Investigational Site Number : 1560017, Beijing
  - Investigational Site Number : 1560022, Beijing
  - Investigational Site Number : 1560030, Beijing
  - Investigational Site Number : 1560006, Dongguan
  - Investigational Site Number : 1560007, Guangzhou
  - Investigational Site Number : 1560019, Guiyang
  - Investigational Site Number : 1560023, Hefei
  - Investigational Site Number : 1560002, Nanchang
  - Investigational Site Number : 1560014, Nanjing
  - Investigational Site Number : 1560008, Ningbo
  - Investigational Site Number : 1560031, Ningbo
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560003, Shijiazhuang
  - Investigational Site Number : 1560029, Sichuan
  - Investigational Site Number : 1560011, Taiyuan
  - Investigational Site Number : 1560012, Taiyuan
  - Investigational Site Number : 1560004, Tianjin
  - Investigational Site Number : 1560025, Tianjin
  - Investigational Site Number : 1560009, Wuxi
  - Investigational Site Number : 1560028, Xi'an
  - Investigational Site Number : 1560020, Xiamen
  - Investigational Site Number : 1560024, Xiamen
  - Investigational Site Number : 1560013, Yichang
  - Investigational Site Number : 1560010, Yueyang
  - Investigational Site Number : 1560021, Zhengzhou
- Greece (11):
  - Investigational Site Number : 3000011, Alexandroupoli
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000010, Athens
  - Investigational Site Number : 3000007, Athens
  - Investigational Site Number : 3000004, Athens
  - Investigational Site Number : 3000006, Athens
  - Investigational Site Number : 3000005, Athens
  - Investigational Site Number : 3000002, Ioannina
  - Investigational Site Number : 3000008, N. Efkarpia
  - Investigational Site Number : 3000009, Palaió Fáliro
  - Investigational Site Number : 3000001, Thessaloniki
- Hungary (10):
  - Investigational Site Number : 3480012, Budapest
  - Investigational Site Number : 3480008, Debrecen
  - Investigational Site Number : 3480005, Edelény
  - Investigational Site Number : 3480004, Hajdúnánás
  - Investigational Site Number : 3480011, Monor
  - Investigational Site Number : 3480007, Mosonmagyaróvár
  - Investigational Site Number : 3480003, Püspökladány
  - Investigational Site Number : 3480001, Százhalombatta
  - Investigational Site Number : 3480013, Szekszárd
  - Investigational Site Number : 3480006, Szombathely
- India (16):
  - Investigational Site Number : 3560011, Ahmedabad
  - Investigational Site Number : 3560021, Bengaluru
  - Investigational Site Number : 3560003, Chandigarh
  - Investigational Site Number : 3560008, Coimbatore
  - Investigational Site Number : 3560016, Faridabad
  - Investigational Site Number : 3560001, Jaipur
  - Investigational Site Number : 3560019, Jodhpur
  - Investigational Site Number : 3560002, Kozhikode
  - Investigational Site Number : 3560014, Lucknow
  - Investigational Site Number : 3560006, Mangaluru
  - Investigational Site Number : 3560018, Mysuru
  - Investigational Site Number : 3560009, Nagpur
  - Investigational Site Number : 3560012, Nagpur
  - Investigational Site Number : 3560015, New Delhi
  - Investigational Site Number : 3560020, Pune
  - Investigational Site Number : 3560004, Vadodara
- Ireland (2):
  - Investigational Site Number : 3720001, Wilton, Cork
  - Investigational Site Number : 3720003, Dublin
- Mexico (12):
  - Investigational Site Number : 4840002, Guadalajara, Jalisco
  - Investigational Site Number : 4840012, Chihuahua, Mexico City
  - Investigational Site Number : 4840006, Mexico City, Mexico City
  - Investigational Site Number : 4840013, Oaxaca, Mexico City
  - Investigational Site Number : 4840004, Monterrey, Nuevo León
  - Investigational Site Number : 4840008, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, Monterrey, Nuevo León
  - Investigational Site Number : 4840014, San Juan del Río, Querétaro
  - Investigational Site Number : 4840010, Villahermosa, Tabasco
  - Investigational Site Number : 4840016, Chihuahua City
  - Investigational Site Number : 4840001, Durango
  - Investigational Site Number : 4840003, Veracruz
- Oman (2):
  - Investigational Site Number : 5120002, Muscat
  - Investigational Site Number : 5120001, Muscat
- Peru (3):
  - Investigational Site Number : 6040001, Lima
  - Investigational Site Number : 6040002, Lima
  - Investigational Site Number : 6040003, Piura
- Puerto Rico (3):
  - Cardio Pulmonary Research Center- Site Number : 8400126, Guaynabo
  - FDI Clinical Research- Site Number : 8400121, San Juan
  - University of Puerto Rico - Medical Sciences Campus- Site Number : 8400128, San Juan
- Romania (9):
  - Investigational Site Number : 6420010, Baia Mare
  - Investigational Site Number : 6420005, Bragadiru
  - Investigational Site Number : 6420007, Brasov
  - Investigational Site Number : 6420002, Brasov
  - Investigational Site Number : 6420004, Codlea
  - Investigational Site Number : 6420011, Craiova
  - Investigational Site Number : 6420001, Deva
  - Investigational Site Number : 6420008, Piteşti
  - Investigational Site Number : 6420009, Timișoara
- Investigational Site Number : 6820008, Mecca, Saudi Arabia
- Slovakia (4):
  - Investigational Site Number : 7030003, Levice
  - Investigational Site Number : 7030001, Poprad
  - Investigational Site Number : 7030002, Spišská Nová Ves
  - Investigational Site Number : 7030005, Topoľčany
- South Africa (11):
  - Investigational Site Number : 7100006, Benoni
  - Investigational Site Number : 7100013, Cape Town
  - Investigational Site Number : 7100004, Cape Town
  - Investigational Site Number : 7100001, Cape Town
  - Investigational Site Number : 7100012, Chatsworth
  - Investigational Site Number : 7100003, Durban
  - Investigational Site Number : 7100009, Durban
  - Investigational Site Number : 7100014, Kempton Park
  - Investigational Site Number : 7100002, Pretoria
  - Investigational Site Number : 7100008, Somerset West
  - Investigational Site Number : 7100007, Vereeniging
- South Korea (10):
  - Investigational Site Number : 4100007, Busan, Busan
  - Investigational Site Number : 4100006, Daegu, Daegu
  - Investigational Site Number : 4100008, Wŏnju, Gangwon-do
  - Investigational Site Number : 4100010, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100009, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul, Seoul-teukbyeolsi
- Taiwan (4):
  - Investigational Site Number : 1580001, Kaohsiung City
  - Investigational Site Number : 1580004, Taichung
  - Investigational Site Number : 1580002, Taipei
  - Investigational Site Number : 1580003, Yunlin
- Turkey (Türkiye) (8):
  - Investigational Site Number : 7920003, Adana
  - Investigational Site Number : 7920007, Ankara
  - Investigational Site Number : 7920008, Ankara
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920006, Izmir
  - Investigational Site Number : 7920009, Kayseri
  - Investigational Site Number : 7920004, Kırıkkale
  - Investigational Site Number : 7920002, Mersin
- United Arab Emirates (2):
  - Investigational Site Number : 7840001, Abu Dhabi
  - Investigational Site Number : 7840002, Abu Dhabi
- United Kingdom (6):
  - Investigational Site Number : 8260004, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260008, Wakefield, Leeds
  - Investigational Site Number : 8260003, Oxford, Oxfordshire
  - Investigational Site Number : 8260002, Bradford
  - Investigational Site Number : 8260005, Liverpool
  - Investigational Site Number : 8260001, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] De Prado Gomez L, Pavord I, Busse W, Brightling CE, Wechsler ME, Rabe KF, Zhang M, Xing J, Jacob-Nara JA, Rowe PJ. Long-term effect of dupilumab on prevention of lung function decline in patients with uncontrolled moderate-to-severe asthma: ATLAS trial design. ERJ Open Res. 2023 Mar 6;9(2):00417-2022. doi: 10.1183/23120541.00417-2022. eCollection 2023 Mar. PMID 36891077
- See also: LPS16676 Asthma clinical study website — https://www.asthmaclinicalstudies.com/?utm_source=ctgov&utm_medium=website
- See also: LPS16676 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25287&tenant=MT_SNY_9011